CLINICAL TRIAL: NCT01049763
Title: Phase I, Open-Label Study to Evaluate Potential Pharmacokinetic of Orally Administered Oseltamivir in Healthy Obese Thai Adult Subjects
Brief Title: Open-Label Pharmacokinetic of Oseltamivir in Healthy Obese Thai Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: South East Asia Infectious Disease Clinical Research Network (Network)
Collaborators: University of Oxford (Other)
Responsible Party: Dr. Podjanee Jittmala, Mahidol-Oxford Tropical Medicine Research Unit Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: SEA 131
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: obese adult; non obese healthy volunteers; oseltamivir carboxylate; pharmacokinetics; healthy volunteers
MeSH Terms: interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regimen A (Experimental): oseltamivir 75 mg single dose
  Interventions: Drug: oseltamivir
- Regimen B (Active Comparator): oseltamivir 150 mg single dose
  Interventions: Drug: oseltamivir

INTERVENTIONS:
Drug: oseltamivir — oseltamivir 150 mg single oral dose oseltamivir 75 mg single oral dose

SUMMARY:
This study is planned to characterize the pharmacokinetic properties of oseltamivir and the active product--oseltamivir carboxylate--in obesity in order to provide clinical guidance for the optimum oseltamivir treatment regimens for severe influenza. It is also a prompt response to a new era influenza plan along with recognition of growing numbers of obese persons.

The study findings will be available for a future management plan in dealing with this virus that is transmitted easily from person to person and has shown substantial antigenic changes over time.

The primary focus of statistical analysis is to verify the effect of obesity on oseltamivir/oseltamivir carboxylate pharmacokinetics as measured by oseltamivir carboxylate Cmax, AUC (0-12), AUC (0-24), C12, λz, and t1/2 and oseltamivir Cmax, AUC (0-12), and C12.

DETAILED DESCRIPTION:
This is an open-label, cross-over, randomized pharmacokinetic study conducted in approximately 12 obese and 12 non obese adult subjects at one study center in Thailand.

Subjects will receive 2 regimens in a random sequence for 2 visits.

1. Regimen A; 75 mg single dose.
2. Regimen B; 150 mg single dose. All dosing will be supervised and documented. Subjects will have 2 hospitalizations to complete visit 2 and visit 3 in their assigned sequence within each. Each visit will require hospitalization for about 40 hours (2 nights and 2 days). The subject will be randomized to receive either regimen A or B on first admission (visit 2). Treatment allocation will be performed using computer-generated list of random permutations of AB sequence.

Subjects who received regimen A will receive regimen B on second admission and vice versa, with more than 3 days wash out period in between. Subjects will return to the study centre for a follow-up visit 7-10 days after completing the last dosing assessments or withdrawing from the study. The total duration of study participation will be approximately 4 weeks from screening through follow-up.

Assessment of the safety profile will be done after each admission by the investigating team before proceeding to the other regimen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as judged by a responsible physician with no abnormality identified on a medical evaluation including medical history and physical examination.
* Males and Females aged between 18 years to 60 years.
* BMI >30 kg/ m2 (BMI = body weight [BW] (kg)/height (m2)) for obese group, BMI 18-24.9 kg/ m2 (BMI = BW (kg)/height (m2)) for control group.
* A female is eligible to enter and participate in this study if she is:

  * of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy
  * or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy
  * or of childbearing potential, has a negative serum pregnancy test at screening and prior to start the study drug in each period, and abstain from sexual intercourse or agrees to using effective contraceptive methods during the study until completion of the follow-up procedures
* A male is eligible to enter and participate in this study if he: agrees to abstain from (or use a condom during) sexual intercourse with females of childbearing potential or lactating females; or is willing to use a condom/spermicide, during the study until completion of the follow-up procedures.
* Read, comprehend, and write at a sufficient level to complete study-related materials.
* Provide a signed and dated written informed consent prior to study participation.
* Normal electrocardiogram (ECG) with QTc <450 msec.
* Willingness and ability to comply with the study protocol for the duration of the trial.

Exclusion Criteria:

* Females who are pregnant, trying to get pregnant, or are lactating.
* The subject has evidence of active substance abuse that may compromise safety, pharmacokinetics, or ability to adhere with protocol instructions.
* A positive pre-study hepatitis B surface antigen, positive hepatitis C antibody, or positive human immunodeficiency virus-1 (HIV-1) antibody result at screening.
* Subjects with a personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de points (heart failure, hypokalemia).
* Subjects with a family history of sudden cardiac death.
* A creatinine clearance <70 mL/min as determined by Cockcroft-Gault equation:

CLcr (mL/min) = (140 - age) * Wt / (72 * Scr) (multiply answer by 0.85 for females). Where age is in years, weight (wt) is in kg, and serum creatinine (Scr) is in units of mg/dL [Cockcroft, 1976].

* History of alcohol or substance abuse or dependence within 6 months of the study: History of regular alcohol consumption averaging >7 drinks/wk for women or >14 drinks/wk for men. One drink is equivalent to 12 g alcohol = 5 oz (150 mL) of wine or 12 oz (360 mL) of beer or 1.5 oz (45 mL) of 80 proof distilled spirits within 6 months of screening.
* Use of prescription or non-prescription drugs except paracetamol at doses of up to 2 grams/day, including vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure.
* Use of live attenuated influenza vaccine, inactivated influenza vaccine, or any other antiinfluenza antiviral medications within 14 days prior to the first dose of investigational product.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
* The subject is unwilling to abstain from ingesting alcohol within 48 hours prior to the first dose of study medication until collection of the final pharmacokinetic sample during each regimen.
* Subjects who have donated blood to the extent that participation in the study would result in more than 300 mL blood donated within a 30-day period.
* Subjects who have a history of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the trial. In addition, if heparin is used during pharmacokinetic sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Subjects with unstable medical conditions that, in the opinion of the investigator would compromise their participation in the trial
* Those who, in the opinion of the investigator, have a risk of non-compliance with study procedures.
* Lack of suitability for participation in this study, for any reason, in the opinion of the investigator.
* AST or ALT >1.5 upper limit of normal (ULN)
* Subjects with history of renal disease, hepatic disease, and/or cholecystectomy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Oseltamivir carboxylate maximum concentration (OC Cmax) and area under the concentration curve 0-12h (OC AUC(0-12)) | 12 hours

SECONDARY OUTCOMES:
Oseltamivir maximum concentration at 12 hours (OS C12) Oseltamivir carboxylate area under the concentration curve 0-24 hours AUC(0-24)), concentration at 24 hours (C24), elimination rate constant (OC-λz), and elimination half life (t1/2) | 1 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Podjanee Jittmala, MD, Principal Investigator — Mahidol-Oxford Tropical Medicine Research Unit Faculty of Tropical Medicine, Mahidol University; Sasithon Pukrittayakamee, Professor, Study Chair — Mahidol University; Pratap Singhasivanon, A/Professor, Study Chair — Mahidol University; Nick White, Professor, Study Chair — Mahidol-Oxford Tropical Medicine Research Unit Faculty of Tropical Medicine, Mahidol University Bangkok, Thailand; Nick Day, Professor, Study Chair — Mahidol-Oxford Tropical Medicine Research Unit Faculty of Tropical Medicine, Mahidol University Bangkok, Thailand; Niklas Lindegardh, A/Professor, Study Chair — Clinical Pharmacology Laboratory Faculty of Tropical Medicine, Mahidol University Bangkok, Thailand; Bob Taylor, MD, Study Chair — Mahidol-Oxford Tropical Medicine Research Unit, Faculty of Tropical Medicine, Mahidol University Bangkok, Thailand
Locations (1):
- Mahidol-Oxford Tropical Medicine Research Unit Faculty of Tropical Medicine, Mahidol University Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Ward P, Small I, Smith J, Suter P, Dutkowski R. Oseltamivir (Tamiflu) and its potential for use in the event of an influenza pandemic. J Antimicrob Chemother. 2005 Feb;55 Suppl 1:i5-i21. doi: 10.1093/jac/dki018. PMID 15709056
- [Background] Tran TH, Nguyen TL, Nguyen TD, Luong TS, Pham PM, Nguyen vV, Pham TS, Vo CD, Le TQ, Ngo TT, Dao BK, Le PP, Nguyen TT, Hoang TL, Cao VT, Le TG, Nguyen DT, Le HN, Nguyen KT, Le HS, Le VT, Christiane D, Tran TT, Menno de J, Schultsz C, Cheng P, Lim W, Horby P, Farrar J; World Health Organization International Avian Influenza Investigative Team. Avian influenza A (H5N1) in 10 patients in Vietnam. N Engl J Med. 2004 Mar 18;350(12):1179-88. doi: 10.1056/NEJMoa040419. Epub 2004 Feb 25. PMID 14985470
- [Background] Chotpitayasunondh T, Ungchusak K, Hanshaoworakul W, Chunsuthiwat S, Sawanpanyalert P, Kijphati R, Lochindarat S, Srisan P, Suwan P, Osotthanakorn Y, Anantasetagoon T, Kanjanawasri S, Tanupattarachai S, Weerakul J, Chaiwirattana R, Maneerattanaporn M, Poolsavathitikool R, Chokephaibulkit K, Apisarnthanarak A, Dowell SF. Human disease from influenza A (H5N1), Thailand, 2004. Emerg Infect Dis. 2005 Feb;11(2):201-9. doi: 10.3201/eid1102.041061. PMID 15752436
- [Background] Treanor JJ, Hayden FG, Vrooman PS, Barbarash R, Bettis R, Riff D, Singh S, Kinnersley N, Ward P, Mills RG. Efficacy and safety of the oral neuraminidase inhibitor oseltamivir in treating acute influenza: a randomized controlled trial. US Oral Neuraminidase Study Group. JAMA. 2000 Feb 23;283(8):1016-24. doi: 10.1001/jama.283.8.1016. PMID 10697061
- [Background] Hayden FG, Treanor JJ, Fritz RS, Lobo M, Betts RF, Miller M, Kinnersley N, Mills RG, Ward P, Straus SE. Use of the oral neuraminidase inhibitor oseltamivir in experimental human influenza: randomized controlled trials for prevention and treatment. JAMA. 1999 Oct 6;282(13):1240-6. doi: 10.1001/jama.282.13.1240. PMID 10517426
- [Background] Hayden FG, Atmar RL, Schilling M, Johnson C, Poretz D, Paar D, Huson L, Ward P, Mills RG. Use of the selective oral neuraminidase inhibitor oseltamivir to prevent influenza. N Engl J Med. 1999 Oct 28;341(18):1336-43. doi: 10.1056/NEJM199910283411802. PMID 10536125
- [Background] de Jong MD, Tran TT, Truong HK, Vo MH, Smith GJ, Nguyen VC, Bach VC, Phan TQ, Do QH, Guan Y, Peiris JS, Tran TH, Farrar J. Oseltamivir resistance during treatment of influenza A (H5N1) infection. N Engl J Med. 2005 Dec 22;353(25):2667-72. doi: 10.1056/NEJMoa054512. PMID 16371632
- [Background] Yen HL, Ilyushina NA, Salomon R, Hoffmann E, Webster RG, Govorkova EA. Neuraminidase inhibitor-resistant recombinant A/Vietnam/1203/04 (H5N1) influenza viruses retain their replication efficiency and pathogenicity in vitro and in vivo. J Virol. 2007 Nov;81(22):12418-26. doi: 10.1128/JVI.01067-07. Epub 2007 Sep 12. PMID 17855542
- [Background] Yen HL, Monto AS, Webster RG, Govorkova EA. Virulence may determine the necessary duration and dosage of oseltamivir treatment for highly pathogenic A/Vietnam/1203/04 influenza virus in mice. J Infect Dis. 2005 Aug 15;192(4):665-72. doi: 10.1086/432008. Epub 2005 Jul 15. PMID 16028136
- [Background] Cockshott WP, Thompson GT, Howlett LJ, Seeley ET. Intramuscular or intralipomatous injections? N Engl J Med. 1982 Aug 5;307(6):356-8. doi: 10.1056/NEJM198208053070607. No abstract available. PMID 7088101
- [Background] Ritschel WA, Kaul S. Prediction of apparent volume of distribution in obesity. Methods Find Exp Clin Pharmacol. 1986 Apr;8(4):239-47. PMID 3724300
- [Background] Abernethy DR, Greenblatt DJ. Drug disposition in obese humans. An update. Clin Pharmacokinet. 1986 May-Jun;11(3):199-213. doi: 10.2165/00003088-198611030-00002. PMID 3524955
- [Background] Beckel MH. Factor affecting the storage of drug and other xenobiotics in adipose tissue. Adv Drug Res 1994; 25: 55-86.
- [Background] Benedek IH, Blouin RA, McNamara PJ. Serum protein binding and the role of increased alpha 1-acid glycoprotein in moderately obese male subjects. Br J Clin Pharmacol. 1984 Dec;18(6):941-6. doi: 10.1111/j.1365-2125.1984.tb02567.x. PMID 6529534
- [Background] Caraco Y, Zylber-Katz E, Berry EM, Levy M. Antipyrine disposition in obesity: evidence for negligible effect of obesity on hepatic oxidative metabolism. Eur J Clin Pharmacol. 1995;47(6):525-30. doi: 10.1007/BF00193706. PMID 7768256
- [Background] Stokholm KH, Brochner-Mortensen J, Hoilund-Carlsen PF. Increased glomerular filtration rate and adrenocortical function in obese women. Int J Obes. 1980;4(1):57-63. PMID 7390700
- [Background] Wattanagoon Y, Stepniewska K, Lindegardh N, Pukrittayakamee S, Silachamroon U, Piyaphanee W, Singtoroj T, Hanpithakpong W, Davies G, Tarning J, Pongtavornpinyo W, Fukuda C, Singhasivanon P, Day NP, White NJ. Pharmacokinetics of high-dose oseltamivir in healthy volunteers. Antimicrob Agents Chemother. 2009 Mar;53(3):945-52. doi: 10.1128/AAC.00588-08. Epub 2008 Dec 22. PMID 19104028
- [Background] Massarella JW, He GZ, Dorr A, Nieforth K, Ward P, Brown A. The pharmacokinetics and tolerability of the oral neuraminidase inhibitor oseltamivir (Ro 64-0796/GS4104) in healthy adult and elderly volunteers. J Clin Pharmacol. 2000 Aug;40(8):836-43. doi: 10.1177/00912700022009567. PMID 10934667
- [Derived] Jittamala P, Pukrittayakamee S, Tarning J, Lindegardh N, Hanpithakpong W, Taylor WR, Lawpoolsri S, Charunwattana P, Panapipat S, White NJ, Day NP. Pharmacokinetics of orally administered oseltamivir in healthy obese and nonobese Thai subjects. Antimicrob Agents Chemother. 2014;58(3):1615-21. doi: 10.1128/AAC.01786-13. Epub 2013 Dec 23. PMID 24366750